CLINICAL TRIAL: NCT07069660
Title: Compass 3: A Novel Transition Program to Reduce Disability After a Stroke
Brief Title: Compass 3: A Novel Transition Program to Reduce Disability After Stroke
Acronym: COMPASS 3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202501232; 2R01HD092398-06A1 (NIH)
Record Dates: First submitted 2025-07-14; First posted 2025-07-17 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Stroke
Keywords: occupational therapy; stroke; adults; environmental modifications
MeSH Terms: conditions — Stroke | interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COMPASS intervention (Experimental): COMPASS is a complex intervention that combines 2 evidence-based treatment strategies at a new point of care (transition from inpatient rehabilitation). The objective of home visits by an occupational therapy (OT) practitioner is to remediate barriers in the home and community that influence daily activities and community participation.
  Interventions: Behavioral: COMPASS
- Education Program (Sham Comparator): A research team member will deliver the program in accordance with "Evidence-Based Educational Guidelines for Stroke Survivors after Discharge Home." Topics may include stroke symptoms, risk factors and preventing stroke recurrence.
  Interventions: Behavioral: Education Program

INTERVENTIONS:
Behavioral: COMPASS — The data from the baseline assessment will be used to develop an environmental modification intervention plan. Environmental modifications will be installed before discharge if possible. Problem areas addressed are participant specific (tailored), but the process to identify and address the target area is systematic. All participants will receive identical intervention components. The standardized components include assessment, identification of problematic activities (and environmental barriers), identification of solutions for each problem, implementation of solution set selected by the participant, training, and active practice of daily activities in one's own home and community.
  Arms: COMPASS intervention
Behavioral: Education Program — The control group will experience the same effects of time and attention in the home but no effect on the outcome of interest.
  Arms: Education Program

SUMMARY:
This study evaluates a program designed to help individuals transition from inpatient rehabilitation to home following an ischemic or hemorrhagic stroke. Half of the participants will receive a stroke education program while the other half will receive an environmental modifications program.

DETAILED DESCRIPTION:
A gap in care exists at the point of transition from inpatient rehabilitation (IR) to home, when survivors encounter new environmental barriers due to the cognitive and sensorimotor sequelae of stroke. Resolving these barriers and improving independence in the community have potential to significantly improve stroke survivors' long-term morbidity.

Investigators will conduct a randomized, controlled multi-center trial (RCT) and concurrent implementation evaluation and review of process data to examine therapeutic efficacy, cost-effectiveness and implementation potential of a compensatory intervention (COMPASS) designed to improve daily activity performance and participation outcomes in persons transitioning home from inpatient rehabilitation (IR) following a stroke.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥55 years at the time of screening
* Acute stroke diagnosis (IS or ICH) verified by the stroke team or medical record
* Independent in activities of daily living (ADLs) prior to stroke (premorbid Modified Rankin Scale score ≤2)
* Plan to discharge to home from an IR
* Capable of giving informed consent which includes compliance with the requirements and duration of participation as listed in the Informed Consent Form (ICF).

Exclusion Criteria:

* Life expectancy <6 months
* Cognitive impairment that the participant's stroke team or a research team member believes impairs their ability to provide informed consent or make reasoned choice including the interpretation of the self-rated scales
* Any communication problem that would prevent study completion
* Residence in a congregate living facility
* Not eligible for a therapeutic pass
* Residence outside of the designated catchment area (specific catchment distance to be determined by each site)
* Site investigator's judgment that the participant would not be able to complete research procedures or interventions
* Participation in another research study that in the site investigator's judgment could interfere or conflict with this research study's assessments or interventions

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2030-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Admission to SNF (skilled nursing facility) | From enrollment to 12 months post-discharge from inpatient rehabilitation facility
  Date and days of admission to a skilled nursing facility

CONTACTS AND LOCATIONS:
Overall Officials: Susan Stark, PhD, Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - University of Missouri, Columbia, Missouri
  - Washington University in St. Louis, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: Yes
Final de-identified data will be preserved and shared with the public via WashU Research Data, an institutional repository managed by the Washington University in St. Louis Libraries. Datasets submitted to the data repository undergo curation prior to publication to ensure that the data are functioning, in the appropriate format, and well documented to facilitate long-term FAIRness (findable, accessible, interoperable and reusable). Submissions receive digital object identifiers minted with DataCite, and the library will retain the deposits for a minimum of 10 years.